CLINICAL TRIAL: NCT03962166
Title: Characterizing Patients With Post-operative Atrial Fibrillation in Relation to Cardiac Surgery by Signal Processed Surface Electrocardiogram (wavECG) and Transthoracic Echocardiography A LAACS-2 Sub-study
Brief Title: Characterizing Patients With POAF in Relation to Cardiac Surgery by wavECG and TTE
Status: Active, not recruiting | Type: Observational
Sponsor: Helena DOMINGUEZ (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Helena DOMINGUEZ, MD, PhD, associate professor, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Other Study IDs: H-17033253-S1
Record Dates: First submitted 2019-05-01; First posted 2019-05-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Left Ventricular Diastolic Dysfunction
Keywords: atrial fibrillation; left ventricular diastolic dysfunction; electrocardiogram; signal processed surface ECG; wavECG; transthoracic echocardiography
MeSH Terms: conditions — Atrial Fibrillation; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: consecutive adult patients undergoing first-time elective open-heart surgery

SUMMARY:
Post-operative atrial fibrillation (POAF) is frequently observed after open-heart surgery. Despite numerous attempts to predict POAF, it remains a challenge to correctly identify the patients at risk. New technologies are available but not yet in cooperated in clinical guidelines and prediction models. We aim at identifying patients at risk of AF occurrence/recurrence after open-heart surgery by use of signal processed surface ECG (wavECG).

The study is an explorative, prospective cohort study of 100 patients undergoing first-time elective open-heart surgery in the Left Atrial Appendage Closure by Surgery-2 (LAACS-2) trial (NCT03724318). Patients are examined by electrocardiogram (ECG), wavECG, transthoracic echocardiography and continuous heart rhythm monitoring. Primary endpoint is occurrence/recurrence of AF. Left ventricular diastolic dysfunction as evaluated by wavECG will be used to predict incidence of primary endpoint.

DETAILED DESCRIPTION:
Introduction: Post-operative atrial fibrillation (POAF) is frequently observed after open-heart surgery,1-3 and atrial fibrillation (AF) is frequently complicated by stroke.4-6 During AF, the electrical activity is uncoordinated and the atrial contraction is reduced, increasing the risk of thrombi formation. Subsequently, the thrombi can enter the general circulation, reach the small intracerebral arteries and block blood flow resulting in ischaemic damage.5,7 Anti-coagulant medicines efficiently prevent ischaemic strokes,8 however many patients are asymptomatic or have vague symptoms why diagnosis can be difficult to obtain.5 Furthermore, AF that occurs secondarily to surgery is currently considered self-limiting and continuous anti-coagulation is not necessarily recommended.4,9 However, cumulating evidence suggest that secondary AF in patients with known heart disease increases the long-term risk of stroke and transitory ischaemic attack, recurrent AF and mortality.10-15 In patients undergoing coronary artery bypass grafting (CABG) new-onset AF is associated with increased long-term risk of stroke and mortality compared to patients without AF.14,15 Though there are well-established risk factors for AF, such as age, arterial hypertension, heart failure, myocardial infarction, heart valve disease and diabetes mellitus, the pathophysiology of AF is complex and not fully understood.6,16,17 Both structural remodelling of the atria and electrical pathways, as well as oxidative stress, calcium overload, myofibroblast activation, microRNAs and inflammation, are mentioned as possible factors involved in initiation and progression of AF.6,16-18 Attempts to create and improve risk stratification models for AF and stroke has previously been done, both in community based cohorts and patients undergoing cardiac surgery, e.g. CHA2DS2-VASC, FHS AF risk score, ARIC risk prediction tool, CHARGE-AF risk model, HAVOC score, SYNTAX score, POAF score and POAF prediction model.19-27 However, it remains challenging to accurately predict occurrence of AF both perioperatively and in the subsequent years.28,29

A recent systematic review and meta-analysis concluded that p-wave terminal force in lead V1 (PTFV1), p-wave duration and maximum p-wave area, are all correlated with stroke,30 and a recent review similarly suggest that short and prolonged p-wave and PTFV1 is correlated with AF.31 sp-ECG by Myovista (Southlake, Texas, USA) is a novel advanced ECG utilizing continues wavelet transform signal processing and can detect left ventricular diastolic dysfunction (LVDD) which is associated with AF and post-operative heart failure in other studies.17,32-35 LA strain and E/LA strain indices predicted new cardiovascular events including strokes, in a stroke population36 In patients undergoing catheter ablation for AF, LA strain can identify patients at risk of AF recurrence37,38 POAF has furthermore been predicted in a cohort of patients with severe aortic stenosis by LA strain indexes.39

Aim: We aim at characterizing patients with AF occurrence by novel, easy, and accessible methods such as electrocardiogram (ECG), signal processed surface ECG (Myovista, wavECG) and transthoracic echocardiography (TTE).

Methods: Explorative, prospective cohort study of adult patients undergoing first-time elective open-heart surgery at Department of Cardiothoracic Surgery at Copenhagen University Hospital, Rigshospitalet. One hundred consecutive patients enrolled in the Left Atrial Appendage Closure by Surgery-2 (LAACS-2) trial (NCT03724318) fulfilling the inclusion/exclusion criteria are included in the current study.

The study is approved by the Regional Committee on Health Research Ethics and all procedures followed are in accordance with the ethical standards of the responsible committee on human experimentation and with the Helsinki Declaration. All patients have signed informed consent prior to study enrolment.

Study timeline: One day prior to surgery; patient charts are reviewed, and ECG, wavECG and TTE are obtained. Anaesthesiologists will report AF occurred during intra-operative cardiac monitoring. Post-surgery cardiac rhythm monitoring is applied for at least 48 hours. At discharge patient charts and monitoring are reviewed for any occurrence of new-onset AF. Three months after surgery, patient charts are reviewed, and patients are invited for a single visit at Department of Cardiology at Frederiksberg hospital, where a control ECG, wavECG and TTE are performed. Deviation of the examination programme is accepted, i.e. patients can decline parts of the pre- or post-surgery examinations and remain in the study for follow-up.

Statistics: Precise sample size calculations are not applicable in this explorative study with LVDD in sp-ECG as primary end-point. One previous study has been performed where wavECG identified patients with LVDD in a population (n=188) referred for computed tomography coronary angiography.32 LA strain measured by TTE predicted POAF in 26 of 60 patients undergoing open-heart surgery for severe aortic stenosis.39 P-wave indices from pre-operative ECGs have predicted POAF in a population of 105 cardiac surgery patients.40 The study will include 100 consecutive patients undergoing open-heart surgery. Expected distribution of patients are n=10 for pre-surgery AF (corresponding to the incidence in the background population 1%6), POAF n= 35-50 (corresponding to the incidence in previous cardiac surgery populations; 35-50%1-3), and non-AF n=40-55 (remaining population). Follow-up will be three months.

Parametric statistics is used as normal distribution is expected (e.g. two-sample unpaired Student's t-test) and data is presented with mean ± standard deviation. All tests are two-sided and a P-value < 0.05 is considered statistically significant. IBM SPSS version 22 will be used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* First time open-heart surgery
* Coronary artery bypass grafting and/or valve surgery
* Signed informed consent

Exclusion Criteria:

* Planned closure of the left atrial appendage
* Planned ablation for atrial fibrillation during surgery
* Ongoing inflammation or infection (including endocarditis)
* Connective tissue disease
* Ongoing cancer (not control)
* Pregnancy
* Follow-up not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients undergoing first-time elective open-heart surgery at Department of Cardiothoracic Surgery at Copenhagen University Hospital not fulfilling any exclusion criteria and who have signed informed consent
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | before discharge within two weeks after surgery
  Occurence/recurrence of atrial fibrillation

OTHER OUTCOMES:
Left atrial dysfunction | Two years post surgery
  Evaluated by speckle-tracking and strain analysis (transthoracic echocardiography)
Left ventricular diastolic dysfunction | Two years post surgery
  Evaluated by wavECG

CONTACTS AND LOCATIONS:
Overall Officials: Helena Dominguez, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Cardiology department Y, Bispebjerg-Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual patient data for primary and secondary outcomes measures will be made available upon reasonable request.

REFERENCES:
- [Result] Ahlsson A, Fengsrud E, Bodin L, Englund A. Postoperative atrial fibrillation in patients undergoing aortocoronary bypass surgery carries an eightfold risk of future atrial fibrillation and a doubled cardiovascular mortality. Eur J Cardiothorac Surg. 2010 Jun;37(6):1353-9. doi: 10.1016/j.ejcts.2009.12.033. PMID 20138531
- [Result] Pillarisetti J, Patel A, Bommana S, Guda R, Falbe J, Zorn GT, Muehlebach G, Vacek J, Sue Min Lai, Lakkireddy D. Atrial fibrillation following open heart surgery: long-term incidence and prognosis. J Interv Card Electrophysiol. 2014 Jan;39(1):69-75. doi: 10.1007/s10840-013-9830-6. Epub 2013 Nov 29. PMID 24293173
- [Result] Lee SH, Kang DR, Uhm JS, Shim J, Sung JH, Kim JY, Pak HN, Lee MH, Joung B. New-onset atrial fibrillation predicts long-term newly developed atrial fibrillation after coronary artery bypass graft. Am Heart J. 2014 Apr;167(4):593-600.e1. doi: 10.1016/j.ahj.2013.12.010. Epub 2014 Jan 4. PMID 24655710
- [Result] Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH; ESC Committee for Practice Guidelines. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Europace. 2010 Oct;12(10):1360-420. doi: 10.1093/europace/euq350. No abstract available. PMID 20876603
- [Result] Healey JS, Crystal E, Lamy A, Teoh K, Semelhago L, Hohnloser SH, Cybulsky I, Abouzahr L, Sawchuck C, Carroll S, Morillo C, Kleine P, Chu V, Lonn E, Connolly SJ. Left Atrial Appendage Occlusion Study (LAAOS): results of a randomized controlled pilot study of left atrial appendage occlusion during coronary bypass surgery in patients at risk for stroke. Am Heart J. 2005 Aug;150(2):288-93. doi: 10.1016/j.ahj.2004.09.054. PMID 16086933
- [Result] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):e199-267. doi: 10.1161/CIR.0000000000000041. Epub 2014 Mar 28. No abstract available. PMID 24682347
- [Result] Dawson AG, Asopa S, Dunning J. Should patients undergoing cardiac surgery with atrial fibrillation have left atrial appendage exclusion? Interact Cardiovasc Thorac Surg. 2010 Feb;10(2):306-11. doi: 10.1510/icvts.2009.227991. Epub 2009 Nov 26. PMID 19942634
- [Result] Aguilar MI, Hart R. Oral anticoagulants for preventing stroke in patients with non-valvular atrial fibrillation and no previous history of stroke or transient ischemic attacks. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD001927. doi: 10.1002/14651858.CD001927.pub2. PMID 16034869
- [Result] Frendl G, Sodickson AC, Chung MK, Waldo AL, Gersh BJ, Tisdale JE, Calkins H, Aranki S, Kaneko T, Cassivi S, Smith SC Jr, Darbar D, Wee JO, Waddell TK, Amar D, Adler D; American Association for Thoracic Surgery. 2014 AATS guidelines for the prevention and management of perioperative atrial fibrillation and flutter for thoracic surgical procedures. J Thorac Cardiovasc Surg. 2014 Sep;148(3):e153-93. doi: 10.1016/j.jtcvs.2014.06.036. Epub 2014 Jun 30. No abstract available. PMID 25129609
- [Result] Siu CW, Jim MH, Ho HH, Miu R, Lee SW, Lau CP, Tse HF. Transient atrial fibrillation complicating acute inferior myocardial infarction: implications for future risk of ischemic stroke. Chest. 2007 Jul;132(1):44-9. doi: 10.1378/chest.06-2733. Epub 2007 Mar 30. PMID 17400657
- [Result] Bishara R, Telman G, Bahouth F, Lessick J, Aronson D. Transient atrial fibrillation and risk of stroke after acute myocardial infarction. Thromb Haemost. 2011 Nov;106(5):877-84. doi: 10.1160/TH11-05-0343. Epub 2011 Aug 25. PMID 21866303
- [Result] Zusman O, Amit G, Gilutz H, Zahger D. The significance of new onset atrial fibrillation complicating acute myocardial infarction. Clin Res Cardiol. 2012 Jan;101(1):17-22. doi: 10.1007/s00392-011-0357-5. Epub 2011 Sep 11. PMID 21910032
- [Result] Asanin MR, Vasiljevic ZM, Matic MD, Mrdovic IB, Perunicic JP, Matic DP, Vujisic-Tesic BD, Stankovic SD, Matic DM, Ostojic MC. The long-term risk of stroke in patients with acute myocardial infarction complicated with new-onset atrial fibrillation. Clin Cardiol. 2009 Aug;32(8):467-70. doi: 10.1002/clc.20603. PMID 19685521
- [Result] Kaw R, Hernandez AV, Masood I, Gillinov AM, Saliba W, Blackstone EH. Short- and long-term mortality associated with new-onset atrial fibrillation after coronary artery bypass grafting: a systematic review and meta-analysis. J Thorac Cardiovasc Surg. 2011 May;141(5):1305-12. doi: 10.1016/j.jtcvs.2010.10.040. Epub 2011 Jan 17. PMID 21247589
- [Result] Horwich P, Buth KJ, Legare JF. New onset postoperative atrial fibrillation is associated with a long-term risk for stroke and death following cardiac surgery. J Card Surg. 2013 Jan;28(1):8-13. doi: 10.1111/jocs.12033. Epub 2012 Nov 27. PMID 23186205
- [Result] Kourliouros A, Camm AJ. Does inflammation influence atrial fibrillation recurrence following catheter ablation? Europace. 2009 Feb;11(2):135-7. doi: 10.1093/europace/eun386. No abstract available. PMID 19168493
- [Result] Jalife J, Kaur K. Atrial remodeling, fibrosis, and atrial fibrillation. Trends Cardiovasc Med. 2015 Aug;25(6):475-84. doi: 10.1016/j.tcm.2014.12.015. Epub 2014 Dec 31. PMID 25661032
- [Result] Khaji A, Kowey PR. Update on atrial fibrillation. Trends Cardiovasc Med. 2017 Jan;27(1):14-25. doi: 10.1016/j.tcm.2016.06.007. Epub 2016 Jun 22. PMID 27520496
- [Result] Mariscalco G, Biancari F, Zanobini M, Cottini M, Piffaretti G, Saccocci M, Banach M, Beghi C, Angelini GD. Bedside tool for predicting the risk of postoperative atrial fibrillation after cardiac surgery: the POAF score. J Am Heart Assoc. 2014 Mar 24;3(2):e000752. doi: 10.1161/JAHA.113.000752. PMID 24663335
- [Result] Kwong C, Ling AY, Crawford MH, Zhao SX, Shah NH. A Clinical Score for Predicting Atrial Fibrillation in Patients with Cryptogenic Stroke or Transient Ischemic Attack. Cardiology. 2017;138(3):133-140. doi: 10.1159/000476030. Epub 2017 Jun 28. PMID 28654919
- [Result] Gu J, Andreasen JJ, Melgaard J, Lundbye-Christensen S, Hansen J, Schmidt EB, Thorsteinsson K, Graff C. Preoperative Electrocardiogram Score for Predicting New-Onset Postoperative Atrial Fibrillation in Patients Undergoing Cardiac Surgery. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):69-76. doi: 10.1053/j.jvca.2016.05.036. Epub 2016 May 24. PMID 27554222
- [Result] Lip GYH, Nielsen PB, Skjoth F, Lane DA, Rasmussen LH, Larsen TB. The value of the European society of cardiology guidelines for refining stroke risk stratification in patients with atrial fibrillation categorized as low risk using the anticoagulation and risk factors in atrial fibrillation stroke score: a nationwide cohort study. Chest. 2014 Nov;146(5):1337-1346. doi: 10.1378/chest.14-0533. PMID 25086251
- [Result] Schnabel RB, Yin X, Gona P, Larson MG, Beiser AS, McManus DD, Newton-Cheh C, Lubitz SA, Magnani JW, Ellinor PT, Seshadri S, Wolf PA, Vasan RS, Benjamin EJ, Levy D. 50 year trends in atrial fibrillation prevalence, incidence, risk factors, and mortality in the Framingham Heart Study: a cohort study. Lancet. 2015 Jul 11;386(9989):154-62. doi: 10.1016/S0140-6736(14)61774-8. Epub 2015 May 7. PMID 25960110
- [Result] Schnabel RB, Sullivan LM, Levy D, Pencina MJ, Massaro JM, D'Agostino RB Sr, Newton-Cheh C, Yamamoto JF, Magnani JW, Tadros TM, Kannel WB, Wang TJ, Ellinor PT, Wolf PA, Vasan RS, Benjamin EJ. Development of a risk score for atrial fibrillation (Framingham Heart Study): a community-based cohort study. Lancet. 2009 Feb 28;373(9665):739-45. doi: 10.1016/S0140-6736(09)60443-8. PMID 19249635
- [Result] Alonso A, Krijthe BP, Aspelund T, Stepas KA, Pencina MJ, Moser CB, Sinner MF, Sotoodehnia N, Fontes JD, Janssens AC, Kronmal RA, Magnani JW, Witteman JC, Chamberlain AM, Lubitz SA, Schnabel RB, Agarwal SK, McManus DD, Ellinor PT, Larson MG, Burke GL, Launer LJ, Hofman A, Levy D, Gottdiener JS, Kaab S, Couper D, Harris TB, Soliman EZ, Stricker BH, Gudnason V, Heckbert SR, Benjamin EJ. Simple risk model predicts incidence of atrial fibrillation in a racially and geographically diverse population: the CHARGE-AF consortium. J Am Heart Assoc. 2013 Mar 18;2(2):e000102. doi: 10.1161/JAHA.112.000102. PMID 23537808
- [Result] Chamberlain AM, Agarwal SK, Folsom AR, Soliman EZ, Chambless LE, Crow R, Ambrose M, Alonso A. A clinical risk score for atrial fibrillation in a biracial prospective cohort (from the Atherosclerosis Risk in Communities [ARIC] study). Am J Cardiol. 2011 Jan;107(1):85-91. doi: 10.1016/j.amjcard.2010.08.049. PMID 21146692
- [Result] Gecmen C, Babur Guler G, Erdogan E, Hatipoglu S, Guler E, Yilmaz F, Unkun T, Cap M, Bengi Bakal R, Bayram T, Deniz Acar R, Candan O, Ozdemir N. SYNTAX score predicts postoperative atrial fibrillation in patients undergoing on-pump isolated coronary artery bypass grafting surgery. Anatol J Cardiol. 2016 Sep;16(9):655-61. doi: 10.5152/AnatolJCardiol.2015.6483. Epub 2015 Nov 18. PMID 27488747
- [Result] Szymanski C, Magne J, Fournier A, Rusinaru D, Touati G, Tribouilloy C. Usefulness of preoperative atrial fibrillation to predict outcome and left ventricular dysfunction after valve repair for mitral valve prolapse. Am J Cardiol. 2015 May 15;115(10):1448-53. doi: 10.1016/j.amjcard.2015.02.027. Epub 2015 Feb 18. PMID 25784520
- [Result] Bessissow A, Khan J, Devereaux PJ, Alvarez-Garcia J, Alonso-Coello P. Postoperative atrial fibrillation in non-cardiac and cardiac surgery: an overview. J Thromb Haemost. 2015 Jun;13 Suppl 1:S304-12. doi: 10.1111/jth.12974. PMID 26149040
- [Result] He J, Tse G, Korantzopoulos P, Letsas KP, Ali-Hasan-Al-Saegh S, Kamel H, Li G, Lip GYH, Liu T. P-Wave Indices and Risk of Ischemic Stroke: A Systematic Review and Meta-Analysis. Stroke. 2017 Aug;48(8):2066-2072. doi: 10.1161/STROKEAHA.117.017293. Epub 2017 Jul 5. PMID 28679858
- [Result] German DM, Kabir MM, Dewland TA, Henrikson CA, Tereshchenko LG. Atrial Fibrillation Predictors: Importance of the Electrocardiogram. Ann Noninvasive Electrocardiol. 2016 Jan;21(1):20-9. doi: 10.1111/anec.12321. Epub 2015 Nov 2. PMID 26523405
- [Result] Sengupta PP, Kulkarni H, Narula J. Prediction of Abnormal Myocardial Relaxation From Signal Processed Surface ECG. J Am Coll Cardiol. 2018 Apr 17;71(15):1650-1660. doi: 10.1016/j.jacc.2018.02.024. PMID 29650121
- [Result] Brecher O, Gulati H, Roistacher N, Zhang H, Shi W, Thaler HT, Amar D. Preoperative Echocardiographic Indices of Diastolic Dysfunction and Brain Natriuretic Peptide in Predicting Postoperative Atrial Fibrillation After Noncardiac Surgery. Anesth Analg. 2017 Apr;124(4):1099-1104. doi: 10.1213/ANE.0000000000001471. PMID 27918330
- [Result] Sellers D, Srinivas C, Djaiani G. Cardiovascular complications after non-cardiac surgery. Anaesthesia. 2018 Jan;73 Suppl 1:34-42. doi: 10.1111/anae.14138. PMID 29313903
- [Result] Melduni RM, Schaff HV, Lee HC, Gersh BJ, Noseworthy PA, Bailey KR, Ammash NM, Cha SS, Fatema K, Wysokinski WE, Seward JB, Packer DL, Rihal CS, Asirvatham SJ. Impact of Left Atrial Appendage Closure During Cardiac Surgery on the Occurrence of Early Postoperative Atrial Fibrillation, Stroke, and Mortality: A Propensity Score-Matched Analysis of 10 633 Patients. Circulation. 2017 Jan 24;135(4):366-378. doi: 10.1161/CIRCULATIONAHA.116.021952. Epub 2016 Nov 30. PMID 27903589
- [Result] Hsu PC, Lee WH, Chu CY, Lee HH, Lee CS, Yen HW, Lin TH, Voon WC, Lai WT, Sheu SH, Su HM. Prognostic role of left atrial strain and its combination index with transmitral E-wave velocity in patients with atrial fibrillation. Sci Rep. 2016 Feb 1;6:17318. doi: 10.1038/srep17318. PMID 26833057
- [Result] Ma XX, Zhang YL, Hu B, Zhu MR, Jiang WJ, Wang M, Zheng DY, Xue XP. The usefulness of global left atrial strain for predicting atrial fibrillation recurrence after catheter ablation in patients with persistent and paroxysmal atrial fibrillation. Arch Cardiovasc Dis. 2017 Aug-Sep;110(8-9):447-455. doi: 10.1016/j.acvd.2016.11.005. Epub 2017 May 18. PMID 28528995
- [Result] Parwani AS, Morris DA, Blaschke F, Huemer M, Pieske B, Haverkamp W, Boldt LH. Left atrial strain predicts recurrence of atrial arrhythmias after catheter ablation of persistent atrial fibrillation. Open Heart. 2017 Apr 28;4(1):e000572. doi: 10.1136/openhrt-2016-000572. eCollection 2017. PMID 28674624
- [Result] Pernigo M, Canneto B, Betta D, Molinari G, Ribichini F, Zannini G, Vassanelli C, Rossi A. Dyspnea following thoracostomy closure after right pneumonectomy: An uncommon echocardiographic diagnosis and therapeutic approach. Echocardiography. 2017 May;34(5):782-785. doi: 10.1111/echo.13505. Epub 2017 Mar 14. PMID 28295572
- [Result] Materazzo C, Piotti P, Mantovani C, Miceli R, Villani F. Atrial fibrillation after non-cardiac surgery: P-wave characteristics and Holter monitoring in risk assessment. Eur J Cardiothorac Surg. 2007 May;31(5):812-6. doi: 10.1016/j.ejcts.2007.02.007. Epub 2007 Mar 6. PMID 17337197